CLINICAL TRIAL: NCT00496106
Title: Stress, Immunity & Cervical Cancer: Biobehavioral Outcomes of a Randomized Trial
Brief Title: Stress, Immunity and Cervical Cancer: Biobehavioral Outcomes
Acronym: CXR01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Lari Wenzel, Professor of Medicine, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2005-4526; R01CA118136-01A1 (NIH)
Record Dates: First submitted 2007-07-02; First posted 2007-07-04 (Estimated); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Arm (Experimental): 6 telephone counseling sessions
  Interventions: Behavioral: Telephone counseling; Behavioral: Telephone interview
- Usual Care Arm (Active Comparator): 6 telephone counseling sessions
  Interventions: Behavioral: Telephone counseling; Behavioral: Telephone interview

INTERVENTIONS:
Behavioral: Telephone counseling — 6 telephone counseling sessions
Behavioral: Telephone interview — telephone interview

SUMMARY:
The purpose of the study is to:

1. Test the efficacy of psychosocial telephone counseling (PTC) for cervical cancer survivors, compared to usual care.
2. Evaluate the longitudinal immune and neuroendocrine parameters in cervical cancer patients who have received PTC, compared to usual care.
3. Examine the longitudinal relationship between PTC associated modulations of quality of life (QOL) measures and biologic parameters (immune and neuroendocrine).

DETAILED DESCRIPTION:
The incidence and mortality rates for invasive cervical cancer in minority, low-income, and less educated women exceeds that for white, higher income, and better educated women. In southern California the incidence and mortality rates for cervical cancer are nearly twice that of non-Latina white women. Our preliminary work supports and extends the extant literature, noting that quality of life can be significantly disrupted among cervical cancer survivors, with qualitative differences in how Latina women experience cancer survivorship. However, there is a paucity of literature on interventions designed to assist cervical cancer survivors manage illness-specific stress and improve health behaviors. Our current NIH-funded work suggests that a six session psychosocial telephone counseling (PTC) intervention can improve QOL and decrease psychological distress, with accompanying intervention-induced neuroendocrine and immune parameter modulations which may be related to disease endpoints. In primary support of these significant biobehavioral findings, the project herein proposes to accomplish the following Specific Aims:

1. Test the efficacy of PTC for cervical cancer survivors, compared to usual care.
2. Evaluate the longitudinal immune and neuroendocrine parameters in cervical cancer patients who have received PTC, compared to usual care.
3. Examine the longitudinal relationship between PTC associated modulations of QOL measures and biologic parameters (immune and neuroendocrine).

To achieve these aims the investigators will randomize patients ascertained through the two SEER cancer registries to PTC (N=125) or usual care (N=125), stratifying on English or Spanish language preference. Assessments will occur at baseline (9-20 months post diagnosis), and three and nine months post enrollment/baseline. Assessments will include evaluation of QOL (overall QOL, psychological distress, coping, social support, sexual functioning), health behaviors, neuroendocrine parameters dehydroepiandrosterone sulfate, growth hormone [DHEA-S, cortisol, GH] and immunologic parameters (natural killers [NK] cell activity, IL-5, interferon, human papillomavirus (HPV) E6/E7 peptides, IL-15, IL 10). This project has significant public health relevance for an important unstudied cancer survivor population, many of whom are poor and underserved. If effective, an intervention which could improve quality of life (QOL) and health behaviors, and enhance neuroendocrine and immune responses for women with cervical cancer could have significant implications toward disease recurrence or survival.

ELIGIBILITY:
Inclusion Criteria:

* Cervical cancer (stage I, II, or III) patients who have completed definitive treatment at least 2 months earlier and who were diagnosed between 9 and 20 months prior to enrollment.

Exclusion Criteria:

* Stage IV cervical cancer.
* Have undergone previous treatment with biological response modifier or prior immunotherapy within 4 weeks of study enrollment.
* Used investigational drugs within 30 days.
* Were under immune suppression for any reason.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2007-08; Primary Completion 2010-08 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of a multicomponent biobehavioral psychosocial telephone counseling (PTC) intervention for cervical cancer survivors, compared to usual care | 10 years

SECONDARY OUTCOMES:
To evaluate the longitudinal immune and neuroendocrine parameters in cervical cancer patients who have received the PTC intervention, compared to usual care | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Lari B Wenzel, PhD, Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine Medical Center, Orange, California, United States

REFERENCES:
- [Derived] Wenzel L, Osann K, Hsieh S, Tucker JA, Monk BJ, Nelson EL. Psychosocial telephone counseling for survivors of cervical cancer: results of a randomized biobehavioral trial. J Clin Oncol. 2015 Apr 1;33(10):1171-9. doi: 10.1200/JCO.2014.57.4079. Epub 2015 Feb 23. PMID 25713429